CLINICAL TRIAL: NCT01970072
Title: A Placebo- and Midazolam-Controlled, Phase Ia, Single Ascending-Dose Study Evaluating the Safety, Pharmacokinetics, and Pharmacodynamics of Remimazolam Tosylate
Brief Title: A Phase Ⅰa Study of Remimazolam Tosylate in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RMZL-PIa
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Healthy
Keywords: Remimazolam Tosylate; Phase Ⅰ study; Health
MeSH Terms: interventions — 4-methylbenzenesulfonic acid; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (11):
- 1.Remimazolam Tosylate (Experimental): Single IV bolus of Remimazolam Tosylate over 1 minute at 0.01 mg/kg body weight
  Interventions: Drug: Remimazolam Tosylate
- 2.Remimazolam Tosylate (Experimental): Single IV bolus of Remimazolam Tosylate over 1 minute at 0.02 mg/kg body weight
  Interventions: Drug: Remimazolam Tosylate
- 3.Remimazolam Tosylate (Experimental): Single IV bolus of Remimazolam Tosylate over 1 minute at 0.05 mg/kg body weight
  Interventions: Drug: Remimazolam Tosylate
- 4.Remimazolam Tosylate (Experimental): Single IV bolus of Remimazolam Tosylate over 1 minute at 0.075 mg/kg body weight
  Interventions: Drug: Remimazolam Tosylate
- 5.Remimazolam Tosylate (Experimental): Single IV bolus of Remimazolam Tosylate over 1 minute at 0.1 mg/kg body weight
  Interventions: Drug: Remimazolam Tosylate
- 6.Remimazolam Tosylate (Experimental): Single IV bolus of Remimazolam Tosylate over 1 minute at 0.15 mg/kg body weight
  Interventions: Drug: Remimazolam Tosylate
- 7.Remimazolam Tosylate (Experimental): Single IV bolus of Remimazolam Tosylate over 1 minute at 0.2 mg/kg body weight
  Interventions: Drug: Remimazolam Tosylate
- 8.Remimazolam Tosylate (Experimental): Single IV bolus of Remimazolam Tosylate over 1 minute at 0.25 mg/kg body weight
  Interventions: Drug: Remimazolam Tosylate
- 9.Remimazolam Tosylate (Experimental): Single IV bolus of Remimazolam Tosylate over 1 minute at 0.3mg/kg body weight
  Interventions: Drug: Remimazolam Tosylate
- 10.Remimazolam Tosylate (Experimental): Single IV bolus of Remimazolam Tosylate over 1 minute at 0.35 mg/kg body weight
  Interventions: Drug: Remimazolam Tosylate
- 11.Midazolam (Active Comparator): Single IV bolus of Midazolam over 1 minute at 0.075 mg/kg body weight
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Remimazolam Tosylate
  Arms: 1.Remimazolam Tosylate; 10.Remimazolam Tosylate; 2.Remimazolam Tosylate; 3.Remimazolam Tosylate; 4.Remimazolam Tosylate; 5.Remimazolam Tosylate; 6.Remimazolam Tosylate; 7.Remimazolam Tosylate; 8.Remimazolam Tosylate; 9.Remimazolam Tosylate
Drug: Midazolam
  Arms: 11.Midazolam

SUMMARY:
The purpose of this study is to evaluate and compare the Pharmacokinetics/Pharmacodynamics and safety of Remimazolam Tosylate with midazolam in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females
* Weight range 50 to 100 kg inclusive
* Body mass index (BMI) 18 to 26 kg/m2

Exclusion Criteria:

* Has a known sensitivity to benzodiazepines, flumazenil, or anesthetic agents, or a medical condition such that these agents are contraindicated
* With evidence of uncontrolled renal, hepatic, central nervous system, respiratory, cardiovascular, or metabolic dysfunction, in the opinion of the investigator or medical monitor
* Has known or suspected history of alcoholism or drug abuse or misuse within 6 months of Screening or evidence of tolerance or physical dependence before dosing with study drug
* With a history of laboratory results that show the presence of hepatitis B surface antigen (HBs Ag), hepatitis C antibody (HCV Ab), or human immunodeficiency virus (HIV)
* Pregnant,lactating
* Mallampati score ≥3

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2013-10-14 (Actual); Primary Completion 2014-06-20 (Actual); Study Completion 2014-06-20 (Actual)

PRIMARY OUTCOMES:
To study the Pharmacokinetics of Remimazolam Tosylate by assessment of drug concentration through blood sample analysis | Pre-dose to 8 hours post-dosee
Bispectral index (BIS) and Modified Observer's Assessment of Alertness/Sedation(MOAA/S) score assessments | Pre-dose to 2 hours post-dose
Adverse event；Vital sign；Physical examination；Laboratory examination；ECG；The nervous system function test | Pre-dose to 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Bei Hu, Professor, Principal Investigator — Peiking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

REFERENCES:
- [Derived] Chen X, Sang N, Song K, Zhong W, Wang H, Jiang J, Huang Y, Hu P. Psychomotor Recovery Following Remimazolam-induced Sedation and the Effectiveness of Flumazenil as an Antidote. Clin Ther. 2020 Apr;42(4):614-624. doi: 10.1016/j.clinthera.2020.02.006. Epub 2020 Mar 13. PMID 32178858
- [Derived] Zhou Y, Hu P, Huang Y, Nuoer S, Song K, Wang H, Wen J, Jiang J, Chen X. Population Pharmacokinetic/Pharmacodynamic Model-Guided Dosing Optimization of a Novel Sedative HR7056 in Chinese Healthy Subjects. Front Pharmacol. 2018 Nov 19;9:1316. doi: 10.3389/fphar.2018.01316. eCollection 2018. PMID 30510509